CLINICAL TRIAL: NCT05617937
Title: Examining the Effects of Connective Tissue Massage on Pain After Thoracotomy - Randomized Controlled Trial
Brief Title: Effects of Connective Tissue Massage on Pain After Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Neriman Temel Aksu, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AkdenizUniversitythoracic
Record Dates: First submitted 2021-03-23; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pain
Keywords: Connective tissue massage; Thoracotomy; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue massage gruop (Experimental): In addition, a total of 5 sessions of connective tissue massage were applied to the experimental group as 1 session a day on the postoperative 1st day, 2nd day, 3rd day, 4th day, 5th day. Connective tissue massage was only performed to the patients in the experimental group. A total of 5 sessions of connective tissue massage were applied to the experimental group as 1 session a day on the postoperative 1st day, 2nd day, 3rd day, 4th day, 5th day. Depending on the area of procedure, each session varied between 15 minutes and 20 minutes.
  Interventions: Other: Massage
- Conventional Physiotherapy and Rehabilitation Group (No Intervention): Standard medical treatment, care and pulmonary rehabilitation program were applied to bonventional Physiotherapy and Rehabilitation Group.The patients were mobilized as early as possible. Starting on the postoperative zeroth day, a postoperative rehabilitation program including pulmonary rehabilitation and early mobilization was applied to every patient in the control and experimental groups by a therapist for 1 week as in routine

INTERVENTIONS:
Other: Massage — The connective tissue massage was started from the lumbosacral region (baseline) and was applied to the lower thoracic, scapular, inter-scapular and cervico-occipital region according to the vascular response of the connective tissue.
  Arms: Connective tissue massage gruop

SUMMARY:
Pain can be quite severe after thoracic surgery and effective pain control is highly effective in preventing secretion accumulation, atelectasis, infection and hypoxemia. The objective was evaluate the effect of a connective tissue massage on pain, applied analgesic amounts and length of hospitalization of the patients.The study was conducted at a thoracic surgery department of university hospital in Turkey. Fifty-four patients with operated by the posterolateral thoracotomy method participated.The patients were randomly allocated to 1 of 2 groups: a control group (n27) and the experimental group (n27). Standard medical treatment, care and pulmonary rehabilitation program were applied to both groups. In addition, a total of 5 sessions of connective tissue massage were applied to the experimental group. Pain level of the patients was evaluated at every 24 hours as of the zeroth postoperative day. VAS was used as a one-dimensional scale for pain assessment. Totally applied analgesic amounts and length of hospitalization of the patients were recorded.

DETAILED DESCRIPTION:
The patients were randomly divided into two groups as the control group and the experimental group by using the Microsoft Excel program (Microsoft Inc., Redmond, WA, USA). The population of the study consisted of the patients who were hospitalized at Thoracic Surgery Clinic and operated by the posterolateral thoracotomy method. The first group of the study consisted of the patients in the control group and the second group consisted of the connective tissue massage group. Lobectomy, pneumonectomy, segmentectomy or wedge resection surgeries were performed together with posterolateral thoracotomy in both patient groups.

Standard medical treatment, care and pulmonary rehabilitation program were applied to both groups. The patients were mobilized as early as possible. Starting on the postoperative zeroth day, a postoperative rehabilitation program including pulmonary rehabilitation and early mobilization was applied to every patient in the control and experimental groups by a therapist for 1 week as in routine.

In addition, a total of 5 sessions of connective tissue massage were applied to the experimental group as 1 session a day on the postoperative 1st day, 2nd day, 3rd day, 4th day, 5th day. Connective tissue massage was only performed to the patients in the experimental group. The procedure was performed while the patient was in the sitting position on a chair. In order to provide relaxation in the connective tissue, the patient was asked to perform a slight anterior tilt and to hold his back upright. The middle fingers were used bilaterally in order to provide traction between the cutaneous tissues. In order to prevent contraindication, the procedure was applied to the tissues that were 2 inch away from the surgical site. Throughout the procedure, oxygen saturation of the patient, if required, the heart rate and blood pressure were followed up. The connective tissue massage was started from the lumbosacral region (baseline) and was applied to the lower thoracic, scapular, inter-scapular and cervico-occipital region according to the vascular response of the connective tissue. A total of 5 sessions of connective tissue massage were applied to the experimental group as 1 session a day on the postoperative 1st day, 2nd day, 3rd day, 4th day, 5th day. Depending on the area of procedure, each session varied between 15 minutes and 20 minutes. On postoperative 0th day, 1st day, 2nd day, 3rd day, 4th day, 5th day, 6th day and 7th day (before the massage in the experimental group) (between 8.00 and 9.00 in the morning); in other words, pain level of the patients (n=54) was evaluated at every 24 hours as of the zeroth postoperative day.

Totally applied analgesic amounts of the patients were recorded on the postoperative 0th day, 1st day, 2nd day, 3rd day, 4th day, 5th day, 6th day, and 7th day. In addition, length of hospitalization of the patients was recorded.In the present study, it was found that the patients with prolonged hospitalization period had higher postoperative pain and the duration of hospitalization was longer in the control group. It was thought that this difference was caused by the effects of connective tissue massage on pain.

ELIGIBILITY:
Inclusion Criteria:

* Applying to Thoracic Surgery Department of Akdeniz University Hospital and undergoing thoracotomy via posterolateral thoracotomy incision,
* Being in age range of 20-75 years,
* Being stable in terms of hemodynamics,
* Having no metastatic dissemination,
* Having no known cerebrovascular disease,
* Having no morbid obesity and heart disease that may inhibit the study,
* Having no cognitive impairment that may inhibit communication,
* Having no previous stroke and the associated influence,
* Having no inconvenience for connective tissue massage as a result of the evaluation made by the physician,
* Agreeing to participate in the study.

Exclusion Criteria:

* Having cardiovascular diseases,

  * Having stage 3 (severe) or stage 4 (very severe) chronic obstructive pulmonary disease (COPD),
  * Having more than 200 cc bleeding per hour from the drainage tubes,
  * Having an intubation period longer than 24 hours,
  * Interventions having a negative effect on the pain such as decortication, diaphragm eventration, thoracic wall resection that are performed by thoracotomy were excluded from in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change of Pain Score | Change from Baseline Pain Score at 7 days.
  On postoperative 0th day, 1st day, 2nd day, 3rd day, 4th day, 5th day, 6th day and 7th day (before the massage in the experimental group) (between 8.00 and 9.00 in the morning); in other words, pain level of the patients (n=54) was evaluated at every 24 hours as of the zeroth postoperative day.
Change of applied analgesic amounts of the patients | Change from Baseline applied analgesic amounts of the patients at 7 days.
  Totally applied analgesic amounts of the patients were recorded on the postoperative 0th day, 1st day, 2nd day, 3rd day, 4th day, 5th day, 6th day, and 7th day. In addition, length of hospitalization of the patients was recorded.

SECONDARY OUTCOMES:
Height in Meters | Initial assessment before surgery.
  The height of all subjects in meters (m) will be noted before the surgery.
Weight in Kilograms | Initial assessment before surgery.
  The weight of all subjects in kilograms (kg) will be noted before the surgery.
Body Mass Index (BMI) in kg/m^2 | Initial assessment before surgery.
  Body Mass Index (BMI) will be calculated with the formula weight (kg)/height (m)^2.

CONTACTS AND LOCATIONS:
Overall Officials: Neriman Aksu, Principal Investigator — Akdeniz Üniversitesi Antalya Sağlık Yüksekokulu
Locations (1):
- Neriman Temel Aksu, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No